CLINICAL TRIAL: NCT06487143
Title: The Effects of the 3-month Formulation of Triptorelin (TP) Compared to the 1-month Formulation on the Efficacy, Glucose and Lipid Metabolism, and Bone Mineral Density(BMD) in Idiopathic Central Precocious Puberty(ICPP)
Brief Title: Efficacy, Metabolism and BMD of the 3-month TP Compared to the 1-month TP in ICPP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhe Meng,MD, Associate chief physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3-month TP vs 1-month TP
Record Dates: First submitted 2024-06-20; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Central Precocious Puberty
Keywords: Central Precocious Puberty; GnRHa; predicted adult height; metabolism; bone mineral density
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3-month triptorelin (Experimental): Triptorelin pamoate is administered via intramuscular injection once every three months
  Interventions: Drug: Triptorelin pamoate（15mg）
- 1-month triptorelin (Active Comparator): Triptorelin acetate 3.75mg is administered via intramuscular injection once every four weeks.
  Interventions: Drug: Triptorelin acetate （3.75mg）

INTERVENTIONS:
Drug: Triptorelin pamoate（15mg） — Triptorelin pamoate 15mg is administered via intramuscular injection once every three months.
  Arms: 3-month triptorelin
Drug: Triptorelin acetate （3.75mg） — Triptorelin acetate 3.75mg is administered via intramuscular injection once every four weeks.
  Arms: 1-month triptorelin

SUMMARY:
The primary objective of this study is to compare the efficacy of the 3-month formulation and 1-month formulation of triptorelin and to assess the short-term effects of the 3-month formulation of triptorelin on glucose and lipid metabolism, body composition, and bone density in Chinese ICPP patients.

DETAILED DESCRIPTION:
Idiopathic central precocious puberty (CPP) is an important treatable disease causing pubertal growth disorders. Gonadotropin-releasing hormone analogs (GnRHa) are the first-line drugs for treating idiopathic central precocious puberty (ICPP). Currently, the 1-month formulation (3.75mg) is the most widely used in China. The development of long-acting formulations will reduce the number of injections and treatment costs for children, as well as reduce the clinical visit burden. The 3-month formulation of Triptorelin Pamoate (15mg) was approved for use in central precocious puberty in March 2023. At present, there is only one publicly reported small-sample, single-arm clinical study in China, and there are no large-sample, real-world, concurrent controlled clinical study data on the efficacy and safety of the 3-month and 1-month formulations of triptorelin in the treatment of central precocious puberty. In currently reported safety events both domestically and internationally, there are no reports on the effects of the 3-month formulation of triptorelin on patients' glucose and lipid metabolism, body composition, and bone density. Our research team previously observed in a small-sample retrospective study of female patients with ICPP that after 1 year of treatment with the 3-month formulation of GnRHa (11.25mg leuprorelin), it effectively inhibited the hypothalamic-pituitary-gonadal axis and bone age progression, improved predicted adult height, and had no serious safety events. Therefore, based on our previous work, we plan to conduct a large-sample, real-world, concurrent controlled study to evaluate the gonadal axis suppression and predicted adult height benefits of the 3-month formulation of triptorelin compared to the 1-month formulation in patients with central precocious puberty (CPP). Additionally, we will assess the short-term effects of the 3-month formulation of triptorelin on glucose and lipid metabolism, body composition, and bone density in ICPP patients. The study results are expected to provide clinical evidence for the application of the 3-month formulation in the treatment of central precocious puberty in China.

ELIGIBILITY:
Inclusion Criteria:

1. Early appearance of secondary sexual characteristics, specifically breast development in girls before 8 years old or menarche before 10 years old, and testicular enlargement in boys before 9 years old.
2. Gonadal enlargement: pelvic ultrasound shows that girls have at least one ovarian follicle with a diameter >4mm, and breast development is at least at Tanner stage II; boys have a testicular volume ≥ 4 ml (measured with Prader orchidometer).
3. GnRH stimulation test: LH peak value ≥ 5 IU/L (chemiluminescence method), with an LH peak/FSH peak ratio ≥ 0.6.
4. Bone age (BA) exceeds chronological age (CA) by 1 year or more (based on bone age assessment during the screening period at this center).
5. Accelerated linear growth, with an annual growth rate higher than that of healthy children of the same age.
6. No prior treatment with gonadotropin-releasing hormone agonists.
7. Body weight of at least 20 kg.

Exclusion Criteria:

1.Target Diseases:

1. Secondary central precocious puberty: This includes central nervous system abnormalities (tumors or space-occupying lesions, acquired injuries, congenital developmental abnormalities, etc.) and other diseases (congenital adrenal hyperplasia, familial male-limited precocious puberty, McCune-Albright syndrome, etc.).
2. Slow-progressing central precocious puberty: Some children show signs of sexual development before the defined age (7-8 years), but the progression of sexual development and bone age is slow, and linear growth remains within the corresponding percentiles.

   2.Treatment History, Medical History, and Concomitant Medical Conditions:
3. Known hypersensitivity to any investigational substance or related compounds.
4. Any chronic disease or treatment deemed by the investigator to potentially interfere with growth or other study endpoints [including but not limited to: long-term glucocorticoid use (excluding short-term topical use), renal failure, diabetes, moderate to severe scoliosis].
5. Girls with a bone age over 12.5 years or menarche ≥ 1 year; boys with a bone age over 14 years (based on bone age assessment during the screening period at this center).
6. Congenital long QT syndrome/12-lead ECG at screening showing QTc ≥ 500 ms corrected by Bazett's formula, excluding other factors causing prolonged QT interval on ECG/12-lead ECG at screening showing QTc between 480 and 499 ms accompanied by unexplained syncope, with no other factors causing prolonged QT interval and no pathogenic mutations.
7. BMI ≥ 95th percentile (same age and gender).

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of LH of ≤ 3 IU/L | 3 months after injection of 3-month TP and 1-month TP
  In the GnRHa stimulation test, triptorelin is administered intravenously at a dose of 0.1 mg/m² (with a maximum dose of 0.1 mg). Blood samples are collected 60 minutes after administration to measure luteinizing hormone (LH) levels.Serum LH levels were measured by electroimmunochemiluminescence assays.

SECONDARY OUTCOMES:
Basal LH（ IU/L),Basal FSH（IU/L), Estradiol (female) (pg/mL)and testosterone (male)(pg/mL) | Month 0, 3 ,6 and 12 after injection of triptorelin 3M and 1M
  Changes in baseline luteinizing hormone (LH) levels ,follicle-stimulating hormone (FSH), estradiol (E2), and testosterone (T) after treatment compared to baseline.Serum LH, FSH, estradiol and testosterone levels were measured by electroimmunochemiluminescence assays.
Tanner stage | Month 0, 3 ,6 and 12 after injection of triptorelin 3M and 1M
  Percentage of children with regression or no progression in Tanner staging. Pubertal stage was determined by an experienced pediatric endocrinologist according to the method proposed by Marshall and Tanner.
Uterine length (female)（mL) and testicular volume (male)(mL) | Month 0, 3 ,6 and 12 after injection of triptorelin 3M and 1M
  Changes in uterine length and ovarian volume for girls, and testicular volume for boys. Pelvic ultrasound will be used to measure the uterine length and ovarian dimensions (length, width, and thickness). The ovarian volume will be calculated using the given formula.The Prader orchidometer will be used to measure the testicular volume before and after treatment.
Growth velocity (cm/y) | Month 0, 3 ,6 and 12 after injection of triptorelin 3M and 1M
  Changes in growth velocity (GV) after treatment compared to baseline.Growth velocity (GV) is typically measured as the annual growth rate, which is the increase in height over a year.
BA/CA | Month 0, 6 and 12 after injection of triptorelin 3M and 1M
  Changes in bone age (BA) and the ratio of bone age to chronological age (BA/CA) compared to baseline. Bone age determination will be conducted using an X-ray imaging device to capture X-ray images of the hand and wrist. The BA will be interpreted using a standardized AI bone age assessment instrument (Yitu system).
PAH(cm) | Month 0, 6 and 12 after injection of triptorelin 3M and 1M
  Predicted adult height (PAH) was calculated using the average tables from the Bayley-Pinneau method
Body composition | Month 0 and 12 after injection of triptorelin 3M and 1M
  Comparison of body fat percentage after treatment to baseline using Dual-Energy X-ray Absorptiometry (DXA).
Bone Mineral Density | Month 0 and 12 after injection of triptorelin 3M and 1M
  Comparison of the lowest T-score among the lumbar spine (L1-L4), total hip, and femoral neck after treatment to baseline using Dual-Energy X-ray Absorptiometry (DXA).
BMISDS | Month 0, 6 and 12 after injection of triptorelin 3M and 1M
  Standard deviation scores (SDS) of body mass index (BMI) were calculated using the 2005 growth chart for Chinese children and adolescents aged 0-18 years.Changes in BMI SDS after Treatment Compared to Baseline
glucose metabolism | Month 0, 6 and 12 after injection of triptorelin 3M and 1M
  Changes in Fasting Blood Glucose(mmol/L), Fasting Insulin（μU/mL), and HOMA-IR After Treatment Compared to Baseline.HOMA-IR was calculated by (Fasting Insulin(μU/mL)×Fasting Glucose(mmol/L)) minus 22.5.
lipid metabolism | Month 0, 6 and 12 after injection of triptorelin 3M and 1M
  Changes in Total Cholesterol (TC)(mg/dL) , Low-Density Lipoprotein (LDL) (mg/dL) ,High-Density Lipoprotein (HDL)(mg/dL), Triglycerides (TG) (mg/dL)After Treatment Compared to Baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Meng, master, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Liyang Liang, PhD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Subspecialty Group of Endocrinologic, Hereditary and Metabolic Diseases, the Society of Pediatrics, Chinese Medical Association; Editorial Board, Chinese Journal of Pediatrics. [Expert consensus on the diagnosis and treatment of central precocious puberty(2022)]. Zhonghua Er Ke Za Zhi. 2023 Jan 2;61(1):16-22. doi: 10.3760/cma.j.cn112140-20220802-00693. Chinese. PMID 36594116
- [Result] Cheuiche AV, da Silveira LG, de Paula LCP, Lucena IRS, Silveiro SP. Diagnosis and management of precocious sexual maturation: an updated review. Eur J Pediatr. 2021 Oct;180(10):3073-3087. doi: 10.1007/s00431-021-04022-1. Epub 2021 Mar 21. PMID 33745030
- [Result] Luo X, Zhang C, Yang Y, Xu X, Cheng X, Wei H, Wang L, Huang F, Shi X, Cabri P. Efficacy and Safety of Triptorelin 3-Month Formulation in Chinese Children with Central Precocious Puberty: A Phase 3, Open-Label, Single-Arm Study. Adv Ther. 2023 Oct;40(10):4574-4588. doi: 10.1007/s12325-023-02617-8. Epub 2023 Aug 16. PMID 37584898
- [Result] Bangalore Krishna K, Fuqua JS, Rogol AD, Klein KO, Popovic J, Houk CP, Charmandari E, Lee PA, Freire AV, Ropelato MG, Yazid Jalaludin M, Mbogo J, Kanaka-Gantenbein C, Luo X, Eugster EA, Klein KO, Vogiatzi MG, Reifschneider K, Bamba V, Garcia Rudaz C, Kaplowitz P, Backeljauw P, Allen DB, Palmert MR, Harrington J, Guerra-Junior G, Stanley T, Torres Tamayo M, Miranda Lora AL, Bajpai A, Silverman LA, Miller BS, Dayal A, Horikawa R, Oberfield S, Rogol AD, Tajima T, Popovic J, Witchel SF, Rosenthal SM, Finlayson C, Hannema SE, Castilla-Peon MF, Mericq V, Medina Bravo PG. Use of Gonadotropin-Releasing Hormone Analogs in Children: Update by an International Consortium. Horm Res Paediatr. 2019;91(6):357-372. doi: 10.1159/000501336. Epub 2019 Jul 18. PMID 31319416
- [Result] Durand A, Tauber M, Patel B, Dutailly P. Meta-Analysis of Paediatric Patients with Central Precocious Puberty Treated with Intramuscular Triptorelin 11.25 mg 3-Month Prolonged-Release Formulation . Horm Res Paediatr. 2017;87(4):224-232. doi: 10.1159/000456545. Epub 2017 Mar 23. PMID 28334719
- [Result] Chung LY, Kang E, Nam HK, Rhie YJ, Lee KH. Efficacy of Triptorelin 3-Month Depot Compared to 1-Month Depot for the Treatment of Korean Girls with Central Precocious Puberty in Single Tertiary Center. J Korean Med Sci. 2021 Aug 30;36(34):e219. doi: 10.3346/jkms.2021.36.e219. PMID 34463062
- [Result] Carel JC, Blumberg J, Seymour C, Adamsbaum C, Lahlou N; Triptorelin 3-month CPP Study Group. Three-month sustained-release triptorelin (11.25 mg) in the treatment of central precocious puberty. Eur J Endocrinol. 2006 Jan;154(1):119-24. doi: 10.1530/eje.1.02056. PMID 16382000
- [Result] Huang S, Zhang L, Gao C, Ou H, Hou L, Liu Z, Wang D, Xu Y, Liang L, Meng Z. Efficacy and safety of leuprorelin 3-month depot (11.25 mg) for idiopathic central precocious puberty treatment of Chinese girls: a single-center retrospective study. J Pediatr Endocrinol Metab. 2023 Nov 20;37(1):15-20. doi: 10.1515/jpem-2023-0410. Print 2024 Jan 29. PMID 37975727
- [Result] Ramos CO, Canton APM, Seraphim CE, Faria AG, Tinano FR, Mendonca BB, Latronico AC, Brito VN. Anthropometric, metabolic, and reproductive outcomes of patients with central precocious puberty treated with leuprorelin acetate 3-month depot (11.25 mg). J Pediatr Endocrinol Metab. 2021 Jul 23;34(11):1371-1377. doi: 10.1515/jpem-2021-0142. Print 2021 Nov 25. PMID 34298591

DOCUMENTS (1):
  • Informed Consent Form (2024-06-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT06487143/ICF_000.pdf